CLINICAL TRIAL: NCT04227613
Title: Prospective Study of Cosmetic Outcome and Quality of Life for Women Undergoing Breast Cancer Surgery
Brief Title: Aspects of Breast-conserving Surgery
Status: Completed | Type: Observational
Sponsor: Lund University (Other)
Collaborators: Region Skane (Other)
Responsible Party: Sponsor
Other Study IDs: 2018/827
Record Dates: First submitted 2020-01-09; First posted 2020-01-13 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Breast Neoplasm; Cosmetic Outcome; Quality of Life
Keywords: Humans; prospective studies; breast neoplasms; breast; patient satisfaction; patient reported outcome measures; oncoplastic breast surgery; follow-up studies; mastectomy; quality of life; Sweden
MeSH Terms: conditions — Breast Neoplasms; Patient Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective study of cosmetic outcome and quality of life for women undergoing breast cancer surgery using patient a reported outcome measure (BREAST-Q) and a computer program validated to assess cosmetic outcomes after breast cancer surgery (BCCT.core) at baseline and on 1-year follow-up.

DETAILED DESCRIPTION:
This is a clinical study with the aim to investigate how breast cancer patient's quality of life changes after breast cancer surgery, as well as looking at the cosmetic outcomes for the same patient group. The study is conducted prospectively, with patients being included forward in time when they are diagnosed with breast cancer in Kristianstad hospital, Sweden. The study started in January 2019 and is expected to continue enrollment for two years, with the aim of recruiting 300 patients. The patients fill out a quality of life questionnaire (Breast-Q) at baseline, which is defined as time of diagnosis, and second Breast-Q questionnaire 1-year post surgery. Photos are also taken of the breasts both preoperatively and postoperatively and the photos are assessed by a computer program validated to assess cosmetic outcomes after breast cancer surgery, called BCCT.core, and secondly the cosmetic results of the breasts are evaluated by the surgeon and patient herself on a 10-grade scale. In addition study specific items covering for example psychiatric comorbidity, BMI and smoking are retrieved.

The study hypothesis is that patients undergoing breast cancer surgery overall have a good quality of life 1-year after their diagnosis, especially if they are treated with a surgical approach that takes into account both the best oncological treatment as well as the best surgical technique for cosmetic outcome, so called oncoplastic surgery. The other hypothesis is that cosmetic results will be overall favorable for the group of patients who are operated with breast-conserving techniques, and most favorable in those patients who have undergone oncoplastic surgery. Secondly the study aims to see if there are other patient related variables that affect the quality of life or cosmetic outcome, for example cytostatic treatment, a high body mass index, smoking or psychiatric history prior to diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Women with breast cancer diagnosed in Central Hospital of Kristianstad from 1/1 2019

Exclusion Criteria:

* Patients who lack the ability to read and write Swedish
* Patients that are not able to understand the information given
* Palliative care patients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All women who are diagnosed with breast cancer in Central Hospital of Kristianstad
Sampling Method: Non-Probability Sample
Enrollment: 351 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Quality of life | Change from baseline (time of diagnosis) to 1-year follow-up
  Breast-Q questionnaire to evaluate quality of life and satisfaction with outcome for the patient.Score 0-100, higher score indicates a better outcome. There is also an additional QoL questionnaire at 1-year follow up (EORTC QLQ-C30 and QLQ-BR23).
Cosmetic outcome | Change from baseline (time of diagnosis) to 1-year follow-up
  BCCT.core (breast cancer conservation treatment. cosmetic results) program, together with both surgeon's and patient's score to evaluate cosmetic outcome.
  BCCT.core scores from 1 to 4. 4 is the worse cosmetic outcome. Patients and surgeon will score from 1-10. Higher score indicates a better cosmetic outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Rydén, Prof, Principal Investigator — Lund University; Tor Svensjö, PhD, Principal Investigator — Region Skåne; Kim Gulis, MD, Principal Investigator — Region Skåne / Lund University
Locations (1):
- Central Hospital of Kristianstad, Kristianstad, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gulis K, Ellbrant J, Bendahl PO, Svensjo T, Ryden L. Health-related quality of life by type of breast surgery in women with primary breast cancer: prospective longitudinal cohort study. BJS Open. 2024 May 8;8(3):zrae042. doi: 10.1093/bjsopen/zrae042. PMID 38829692